CLINICAL TRIAL: NCT02989220
Title: A Feasibility and Acceptability Study and a Qualitative Process Evaluation of a Coping Intervention for Women With Recurrent Miscarriage
Brief Title: Feasibility Study of a Coping Intervention for Recurrent Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RHM O&G0207
Record Dates: First submitted 2016-10-14; First posted 2016-12-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Miscarriage
Keywords: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Will receive the PRCI in addition to the current recommended care pathway
  Interventions: Other: Positive Reappraisal Coping Intervention
- Control Group (No Intervention): Will follow the current recommended care pathway

INTERVENTIONS:
Other: Positive Reappraisal Coping Intervention
  Arms: Intervention group

SUMMARY:
Some women experience the pain of miscarriage on numerous occasions. Studies show that these women experience feelings of anxiety and distress during the early stages of a new pregnancy as they worry another miscarriage will occur. This study will investigate whether a coping strategy, developed for a similar group of women, would be acceptable and useful to women suffering recurrent miscarriage, and reduce the anxiety and worry they experience. A secondary aim of the study is to develop a deeper understanding of the experiences and feelings of women in the early stages of a new pregnancy, following multiple miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* Women with three or more miscarriages
* Women aged >18 years
* Willing and able to give written consent

Exclusion Criteria:

* Women will be excluded from this study if they do not speak English well enough to understand and complete study materials. This criterion is in place because the study materials (including PRCI) are not currently available in translation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients finding the proposed methods of recruitment, randomisation, intervention and follow-up acceptable | Through Study Completion - Average of 1 year
  How acceptable are the proposed methods of recruitment, randomisation, intervention and follow-up?
Number of patients recruited into the study using current inclusion/exclusion criteria | Through Study Completion - Average of 1 year
  Is it possible to achieve acceptable recruitment and retention rates within each centre, taking into account defined inclusion/exclusion criteria?
Number of completed questionnaires | Through Study Completion - Average of 1 year
  Are the proposed study questionnaires and data collection methods appropriate?
Data collected from questionnaires | Through Study Completion - Average of 1 year
  Is there a preliminary indication of an effect of the PRCI?

SECONDARY OUTCOMES:
Data Collected from questionnaires | Through Study Completion - Average of 1 year
  Qualitative analysis of questionnaires to explore in-depth women's subjective experience of the study intervention and research methods (including study outcome measures).
Data Collected from questionnaires | Through Study Completion - Average of 1 year
  Qualitative analysis of questionnaires to provide information to refine the study intervention (if required).
Data Collected from questionnaires | Through Study Completion - Average of 1 year
  Qualitative analysis of questionnaires to strengthen further in-depth understanding of the initial experience of pregnancy following repeated miscarriages.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Anne Hospital, Southampton, United Kingdom